CLINICAL TRIAL: NCT02888444
Title: Smoking Relapse Prevention Among COPD Ex-smokers
Acronym: SPACE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Natalie Walker, Associate Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Smoking Cessation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Varenicline plus behavioural support (Active Comparator): 12 weeks extended treatment with varenicline, plus relapse prevention-orientated behavioural support
  Interventions: Drug: Varenicline; Behavioral: Behavioural support
- Placebo plus behavioural support (Placebo Comparator): 12 weeks extended treatment with placebo, plus relapse prevention-orientated behavioural support
  Interventions: Behavioral: Behavioural support; Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Two 0.5mg tablets taken twice daily
  Other Names: Champix
  Arms: Varenicline plus behavioural support
Behavioral: Behavioural support — Consisting of the study-specific doctor delivering relapse prevention orientated behavioural support at the time of consultation, plus six 10-15 minute calls over the 12 weeks delivered by a research assistant.
Drug: Placebo — Two 0.5mg tablets taken twice daily
  Arms: Placebo plus behavioural support

SUMMARY:
A placebo-controlled trial to determine whether recent ex-smokers with COPD who successfully stop smoking after taking varenicline are less likely to relapse back to smoking if they continue using varenicline for a further 12 weeks

DETAILED DESCRIPTION:
Smoking remains the leading cause of Chronic Obstructive Pulmonary Disease (COPD), a leading cause of death and disability in New Zealand. COPD particularly affects indigenous Māori and Pacific people, given their higher rates of smoking. COPD patients tend to have a higher level of nicotine dependence and, as a result, often find quitting harder and are more likely to relapse back to smoking. A clinical trial (N=262) is planned in Auckland, New Zealand to determine whether extended varenicline treatment combined with behavioural support can prevent relapse back to smoking in recent ex-smokers with COPD. Smoking cessation and relapse prevention are the most cost-effective interventions available for COPD patients that smoke, irrespective of their disease stage. The trial has the potential to significantly improve the outcomes of this common and chronic health condition in New Zealand.

ELIGIBILITY:
Inclusion Criteria:

* Daily smokers
* Diagnosed with COPD (as per the Global Initiative for Chronic Obstructive Lung Disease [GOLD] criteria, namely: a characteristic clinical picture of dyspnea, cough or sputum, with a history of exposure to risk factors, plus a post-bronchodilator forced expiratory volume in one second / forced vital capacity FEV1/FVC ratio of <0.70)
* Have stable COPD (i.e. no exacerbation, hospital admission, or use of antibiotics or prednisone in the past six weeks)
* Can provide consent
* Reside in the Auckland region of New Zealand
* Eligible under New Zealand special authority to receive subsidised varenicline
* Prepared to make a quit attempt with varenicline
* Have access to a phone

Exclusion Criteria:

* A history of definite asthma and/or atopy
* Contraindications to varenicline
* Used varenicline in the past 12 months
* A history of serious psychiatric illness or significant cognitive impairment
* Major or uncontrolled co-morbidities (such as uncontrolled heart failure, infection or rapidly progressive condition)
* A life expectancy of < 12 months
* Are currently using another cessation medication (including e-cigarettes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence | 12 weeks post-randomisation
  Continuous (lapse-free) abstinence biochemically validated using a carbon monoxide reading of <10 ppm.

SECONDARY OUTCOMES:
Continuous abstinence | 24 weeks post-randomisation
  Biochemically validated continuous (lapse-free) abstinence
7-day point prevalence abstinence | 12 weeks post-randomisation
  Biochemically validated 7-day point prevalence abstinence, defined as no smoking in the last seven days, not even a puff.
7-day point prevalence abstinence | 24 weeks post-randomisation
  Biochemically validated 7-day point prevalence abstinence, defined as no smoking in the last seven days, not even a puff.
Time to lapse | 12 weeks post-randomisation
  Time to first lapse, defined as time to first cigarette smoked (even a puff)
Time to lapse | 24 weeks post-randomisation
  Time to first lapse, defined as time to first cigarette smoked (even a puff)
Time to relapse | 12 weeks post-randomisation
  Time to first relapse, defined as smoking ≥five cigarettes a day for three consecutive days.
Time to relapse | 24 weeks post-randomisation
  Time to first relapse, defined as smoking ≥five cigarettes a day for three consecutive days.
Cigarettes per day | 12 weeks post-randomisation
  Cigarettes smoked per day, if returned to smoking
Cigarettes per day | 24 weeks post-randomisation
  Cigarettes smoked per day, if returned to smoking
COPD exacerbations requiring hospitalisation | 12 weeks post-randomisation
  The number of COPD exacerbations in the past 12 weeks, defined as a worsening of COPD respiratory symptoms that resulted in a course of antibiotics and/or oral steroids; or an unscheduled visit to GP, urgent care, Emergency Department or as an inpatient. Data will be validated against medical records using data linkage.
COPD exacerbations requiring hospitalisation | 24 weeks post-randomisation
  The number of COPD exacerbations in the past 12 weeks, defined as a worsening of COPD respiratory symptoms that resulted in a course of antibiotics and/or oral steroids; or an unscheduled visit to GP, urgent care, Emergency Department or as an inpatient. Data will be validated against medical records using data linkage.
Urge to smoke/cravings | 12 weeks post-randomisation
  The physical signs and symptoms associated with withdrawal will be measured using the Mood and Physical Symptoms Scale (MPSS).
Urge to smoke/cravings | 24 weeks post-randomisation
  The physical signs and symptoms associated with withdrawal will be measured using the Mood and Physical Symptoms Scale (MPSS).
Cigarette dependence | 12 weeks post-randomisation
  Cigarette dependence, as measured by the Fagerström Test of Cigarette Dependence
Cigarette dependence | 24 weeks post-randomisation
  Cigarette dependence, as measured by the Fagerström Test of Cigarette Dependence
Health-related quality of life | 12 weeks post-randomisation
  Measured using the EQ-5D
Health-related quality of life | 24 weeks post-randomisation
  Measured using the EQ-5D
Serious adverse events | 12 weeks post-randomisation
Serious adverse events | 24 weeks post-randomisation

OTHER OUTCOMES:
Medication adherence (Script redeemed) | 12 weeks post-randomisation
  Question asked about whether they redeemed their allocated script
Question about medication compliance (pill count). | 12 weeks post-randomisation
  Ask about how many of their allocated pills they took
Question about use of other cessation products | 12 weeks post-randomisation
  Questions will be asked about whether other cessation products were used and if so, what type. E-cigarettes will be considered a possible cessation product.
Questions asked about the use of other cessation products | 24 weeks post-randomisation
  Questions will be asked about whether other cessation products were used and if so, what type. E-cigarettes will be considered a possible cessation product.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Walker, PhD, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- National Institute for Health Innovation, University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No